CLINICAL TRIAL: NCT05377164
Title: Long Term Effects of Different Dietary Protocols on Determinants of Health in Patients' Lymphocytes Analysed by FTIR
Brief Title: Long Term Effects of Different Dietary Protocols on Determinants of Health in Patients' Lymphocytes
Acronym: FTIR
Status: Completed | Type: Observational
Sponsor: University of Primorska (Other)
Collaborators: Elettra Synchrotron Trieste (Unknown)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, assoc. prof., University of Primorska
Other Study IDs: DIETE-FTIR
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Asymptomatic Condition
Keywords: diet; lipid peroxidation; DNA damage
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vegetarian group
  Interventions: Behavioral: food choices
- Omnivorous group
  Interventions: Behavioral: food choices
- Low carbohydrate group
  Interventions: Behavioral: food choices

INTERVENTIONS:
Behavioral: food choices — Analysis of lymphocytes isolated from the peripheral blood of participants who had been on vegetarian, ketogenic or normal mixed diet for at least one year will be performed.

SUMMARY:
Food choices and eating habits play an important role in the management of common noncommunicable diseases, i.e. diabetes type II, hypertension, metabolic syndrome and others. However, for many popular diets there is yet no consensus on their actual ability to exert health effects and, regardless of some promising results, the underlying molecular mechanisms are not entirely clear. FTIR analysis could provide interesting new information; we therefore propose the analysis of lymphocytes isolated from the peripheral blood of participants who had been on vegan, ketogenic or normal mixed diet for at least one year. In particular we plan to monitor differences in lipid peroxidation, membrane permeability, protein synthesis and DNA damage. All these parameters are important in the development of the above mentioned diseases and were previously shown to be detectable by FTIR. The results will contribute importantly to the understanding of the long-term effects of the respective lifestyle and will allow the formulation of better dietary recommendations to the public.

DETAILED DESCRIPTION:
Scientific Background: In the overall population there is an increasing awareness that with a healthy lifestyle many chronic non-communicable diseases can be prevented or delayed in their progression. Among them diabetes type II, metabolic syndrome, hypertension and atherosclerosis are recognized as major public health issues also causing the highest proportion of deaths in the modern world. Food choices and eating habits in general play an important role in management of these diseases. There are, however, many popular diets for which there is yet no consensus on their actual possibility to exert health effects. Dietary protocols where whole food groups are excluded are especially known to have some beneficial but also some harmful effects, in particular when not planned properly and used for long periods. Two extremely different lifestyle choices are particularly common in recent years, namely low carbohydrate/high fat (LCHF) diet and vegetarian diet. In the first one, also called ketogenic diet, one eliminates all carbohydrate rich foods, such as fruit, legumes and cereals, but consumes a lot of fats, even up to 90 % of daily energy intake. Such diet is very efficient as a weight-loss program (Mohorko et al., 2019) and when used for shorter periods, was shown to have no adverse effects on total cholesterol or LDL levels. It was also efficient in decreasing the levels of serum glucose and triglycerides (Bueno et al., 2013), but in some cases was calcium deficient (Kenig et al., 2019). Long term effects have not been well investigated and a concern that high fat intake may cause more oxidative stress due to increased beta oxidation remains. Vegan diet, on the other hand, also eliminates a whole food group (meat and dairy products), which may cause depletion of some micronutrients, such as iron and vitamin B12. But, such diet is rich in antioxidants, decreases cholesterol levels and seems to increase longevity (Rizza et al., 2014). Again, studies investigating long-term effects are few.

Motivation for the proposal: In recent years, it has been shown that FTIR can identify many cellular characteristics that are related to the overall "health" of a cell. In the lymphocytes of rats under stress, increased lipid peroxidation was detected by FTIR (Vargas-Caraveo et al., 2014). In human oocytes spectral bands related to lipid saturation, membrane permeability, protein degradation and altered lipid synthesis were found to be changed with aging (Gioacchini et al., 2014). When investigating effects of diets, it is reasonable to expect that lipid content in the cells may change, there may also be differences in the extent of lipid peroxidation or other consequences of oxidative stress. DNA damage, for example, such as single and double strand breaks or DNA-protein cross links, could be induced or inhibited by different dietary ingredients and also identified with FTIR (Sofińska et al., 2020). All these parameters are very important, since increased lipid peroxidation is one of the factors contributing to the development of atherosclerosis, whereas lymphocyte membrane permeabilization and DNA damage are related to cell death and consequential impairment of the immune system. There are studies showing relevant contribution of different diets to these diseases, but underlying molecular mechanisms are not entirely clear. FTIR analysis could then provide interesting novel information, which is the objective of this proposal. In contrast to several biochemical parameters (i.e. cholesterol levels) that somewhat fluctuate depending on recently consumed foods, FTIR analysis of lymphocytes might give information on long-term consequences of a particular lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* 18,5 < BMI < 30 kg/m2
* asymptomatic for any disease
* medication free
* same pattern of eating in the last 3 months
* stable body mass in the last 3 months

Exclusion Criteria:

* BMI < 18,5 and > 30 kg/m2
* presence of any chronic disease
* taking any medications
* changed eating pattern in the last 3 months
* unstable body mass in the last 3 months
* taking antibiotics in the last 3 months

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Asymptomatic adults
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Fourier transform infrared spectra of absorbance at wavelenghts from 500 to 5000 cm-1 | through study completion, an average of 4 months
  Different chemical bonds absorb light at different wavelenghts. This gives information on lipid, protein, DNA, carbohydrate composition of a cell. For individual cells, 256 scans per spectrum will be averaged at 4 cm-1 spectral resolution in transmission mode (15X condenser/objective), 100 cells per sample will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Saša Kenig, PhD, Principal Investigator — University of Primorska Faculty of Health Sciences, Polje 42 SI-6310 Izola
Locations (1):
- University of Primorska Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bueno NB, de Melo IS, de Oliveira SL, da Rocha Ataide T. Very-low-carbohydrate ketogenic diet v. low-fat diet for long-term weight loss: a meta-analysis of randomised controlled trials. Br J Nutr. 2013 Oct;110(7):1178-87. doi: 10.1017/S0007114513000548. Epub 2013 May 7. PMID 23651522
- [Background] Barraza-Garza G, Castillo-Michel H, de la Rosa LA, Martinez-Martinez A, Perez-Leon JA, Cotte M, Alvarez-Parrilla E. Infrared Spectroscopy as a Tool to Study the Antioxidant Activity of Polyphenolic Compounds in Isolated Rat Enterocytes. Oxid Med Cell Longev. 2016;2016:9245150. doi: 10.1155/2016/9245150. Epub 2016 Apr 26. PMID 27213031
- [Background] Gioacchini G, Giorgini E, Vaccari L, Ferraris P, Sabbatini S, Bianchi V, Borini A, Carnevali O. A new approach to evaluate aging effects on human oocytes: Fourier transform infrared imaging spectroscopy study. Fertil Steril. 2014 Jan;101(1):120-7. doi: 10.1016/j.fertnstert.2013.09.012. Epub 2013 Oct 17. PMID 24140036
- [Background] Kenig S, Petelin A, Poklar Vatovec T, Mohorko N, Jenko-Praznikar Z. Assessment of micronutrients in a 12-wk ketogenic diet in obese adults. Nutrition. 2019 Nov-Dec;67-68:110522. doi: 10.1016/j.nut.2019.06.003. Epub 2019 Jun 14. PMID 31445313
- [Background] Mohorko N, Cernelic-Bizjak M, Poklar-Vatovec T, Grom G, Kenig S, Petelin A, Jenko-Praznikar Z. Weight loss, improved physical performance, cognitive function, eating behavior, and metabolic profile in a 12-week ketogenic diet in obese adults. Nutr Res. 2019 Feb;62:64-77. doi: 10.1016/j.nutres.2018.11.007. Epub 2018 Nov 12. PMID 30803508
- [Background] Rizza W, Veronese N, Fontana L. What are the roles of calorie restriction and diet quality in promoting healthy longevity? Ageing Res Rev. 2014 Jan;13:38-45. doi: 10.1016/j.arr.2013.11.002. Epub 2013 Nov 27. PMID 24291541
- [Background] Sofinska K, Wilkosz N, Szymonski M, Lipiec E. Molecular Spectroscopic Markers of DNA Damage. Molecules. 2020 Jan 28;25(3):561. doi: 10.3390/molecules25030561. PMID 32012927
- [Background] Vargas-Caraveo A, Castillo-Michel H, Mejia-Carmona GE, Perez-Ishiwara DG, Cotte M, Martinez-Martinez A. Preliminary studies of the effects of psychological stress on circulating lymphocytes analyzed by synchrotron radiation based-Fourier transform infrared microspectroscopy. Spectrochim Acta A Mol Biomol Spectrosc. 2014 Jul 15;128:141-6. doi: 10.1016/j.saa.2014.02.148. Epub 2014 Mar 12. PMID 24667417